CLINICAL TRIAL: NCT05062135
Title: Abnormalities of the Endometrium Persist Despite Adequate Progesterone Supplementation in the Polycystic Ovary Syndrome
Brief Title: Progesterone Action on Endometrium of PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Edmund Baracat, Full Professor and head of Discipline, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21253613.6.0000.0068
Record Dates: First submitted 2021-09-02; First posted 2021-09-30 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Polycystic Ovary; Progesterone Resistance
Keywords: PCOS; Progesterone; endometrium
MeSH Terms: conditions — Polycystic Ovary Syndrome; Progesterone Resistance | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: A prospective open-label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morphological analysis of endometrium (Experimental): PCOS: Seventeen PCOS subjects underwent two endometrial biopsies after the first P4-treated cycle, the first between days 5-9 of the cycle and the other between days 20-22 (i.e., under P4 treatment) of the cycle.
  Controls: Thirteen ovulatory control women under two endometrial biopsies, performed after the first month of luteal P4 treatment, the first between days 5-9 and the second between days 20-22 of the cycle To quantify the parameters of interest, images were captured using a high-resolution camera (AxioCam-MCR, Carl Zeiss) adapted to a light microscope (Axiolab, Carl Zeiss) and adjusted with 40× objective lenses. The images were transmitted to a computer with AxioVision Rel 4.2 software (Carl Zeiss). For assessment of glandular and surface epithelial thickness, cell count, and counting newly formed blood vessels, ten images of each endometrial sample were made for each patient. For VEGF-C determination, the numerical density of blood vessels per mm2 was established
  Interventions: Drug: Progesterone 400 Mg Vaginal Suppository on PCOS

INTERVENTIONS:
Drug: Progesterone 400 Mg Vaginal Suppository on PCOS — The same drug will be used in control group
  Other Names: Progesterone 400 Mg Vaginal Suppository on control group

SUMMARY:
Objective: To study the influence of metabolic factors on the action of progesterone on the endometrium of women with PCOS.

Design: A prospective open-label clinical trial. Setting: Participants were recruited from an outpatient reproductive endocrinology clinic at an academic tertiary medical care center from 2014 to 2019.

Subjects: To assess the sole effect of progesterone (P4) on the endometrium we studied amenorrheic (cycles> 90 days) women with PCOS (n=23), comparing them to healthy eumenorrheic control women ( n=13).

Intervention(s): All subjects underwent an endometrial biopsy (EB) in the follicular phase of the first study cycle. They were then treated with micronized P4 (400 mg/day x 10 days intravaginally) from days 14-28 of the cycle, and a second EB was performed between days 20-24 of the cycle (second phase).

Main Outcome Measure(s): EB samples were analyzed under light microscopy for histomorphometric analysis.

DETAILED DESCRIPTION:
PATIENTS AND METHODS

Subjects Inclusion criteria for PCOS women will be: a) ages 18 to 35 years, and b) PCOS was defined by the Rotterdam criteria, which includes two of the following three features: a) oligo-amenorrhea; b) clinical or biochemical signs of hyperandrogenism; and c) polycystic ovaries (6). These criteria yield four PCOS phenotypes (A thru D) (1-3). Controls were recruited from the family planning outpatient office. All participants will be healthy women ages 18 to 35 years with regular menstrual cycles, no evidence of hirsutism, no comorbidities, and not using hormone medications in the previous 3 months.

Exclusion criteria are as follows: a) use of any hormone treatment in the previous 3 months; b) other causes of anovulation as evidenced by abnormal levels of prolactin, cortisol, dehydroepiandrosterone sulphate (DHEAS), 17-hydroxyprogesterone (17-OHP), androstenedione, thyroid-stimulating hormone (TSH), and free T4, in blood samples obtained between days 2 and 5 of the cycle in cycling subjects or on any other day in amenorrheic subjects; c) gynecologic disorders or other associated diseases, such as endometriosis, hypertension, or diabetes mellitus; d) follicle-stimulating hormone (FSH) >15 UI/L (cycle days 2-5); or e) a positive β-subunit of human chorionic gonadotropin (β-HCG).

Study Protocol

This trial was previously approved by the Research Ethics Committee (#21253613.6.0000.0068) of the Faculdade de Medicina, Hospital das Clínicas, Universidade de São Paulo (FMUSP), São Paulo, Brazil. The patients will be evaluated at Gynecology Outpatient office. The patients will be divided into two groups: a) PCOS and b) controls. All subjects will be cared for at the Endocrinology Gynecology Section and the Human Reproductive Center of the Gynecology Division, Hospital das Clínicas, FMUSP. After signing the informed consent will be written in accordance with Resolution 196/96 of the National Health Board (Resolução 196/96 do Conselho Nacional de Saúde), all subjects will be included in the study and evaluated as follows:

Preselection: This visit includes the following: interview for medical history; overall physical and gynecologic examinations; weight measurement (scale Filizola, model PL-150, with a capacity for 150 kg); height measurement with a metal stadiometer attached to the scale; abdominal circumference (AC) measurement with a measuring tape at the narrowest region between the last costal arch and the iliac crest; hip circumference (HC) measured around the circumference of hips at the top of the iliac crest and buttocks, body mass index (BMI) and blood pressure (BP) measurement; hirsutism according to the modified Ferriman-Gallwey (mFG) scoring system with nine areas, with patients with a score higher than 8 score deemed hirsute.

The menstrual cycle are considered as normal when the interval between periods was 21 to 35 days, and the blood flow lasted no more than 7 days. The cycle was characterized as anovulatory when the span between blood flows was >35 days (1). Amenorrhea is defined as the absence of a menstrual flow for a period corresponding to the three previous cycles or for >90 days (1,20).

Bloods will be collected and a transvaginal pelvic ultrasound will be performed on all study subjects.

Study A: Six PCOS patients with amenorrhea (cycles >90 days) and negative β-HCG will be prescribed daily micronized P4 (400 mg) administrated via the vaginal route for 10 days. Two endometrial biopsies will be performed, one between the 5th and 9th day and the other between the 21st and 24th day (under the second treatment cycle with P4) of the menstrual cycle (day 1 being the first day of vaginal bleeding). A third biopsy will be repeated on the 4th cycle of P4 treatment, between cycle days 21 and 24 (Fig. 2). This part of the study will be designed to assess whether P4 could transform proliferative into secretory endometrium, regardless of the number of treatment cycles.

Study B:

PCOS: Seventeen PCOS subjects underwent two endometrial biopsies after the first P4-treated cycle, the first between days 5-9 of the cycle and the other between days 20-22 (i.e., under P4 treatment) of the cycle.

Controls: Thirteen ovulatory control women under two endometrial biopsies, will be performed after the first month of luteal P4 treatment, the first between days 5-9 and the second between days 20-22 of the cycle.

Assays The oral glucose tolerance test (OGTT) consisted of 75 grams of glucose administered orally after three days of a carbohydrate-rich diet; blood samples for glucose and insulin measurements were drawn before administration of the glucose solution and 30, 60, 90, and 120 minutes after taking the glucose solution.

Plasma glucose concentration was determined by the glucose oxidase method. All lipid measurements were taken directly in the plasma samples. Total cholesterol and triglycerides were assessed using enzyme methods (Roche Laboratories). The HDL-C was quantified by the same method and LDL-C was estimated with the Friedwald formula. The glycated hemoglobin were measured using high-performance liquid chromatography (with the use of the Tosoh A1c 2.2 Plus Glycohemoglobin Analyzer method in 2003-2004 and the Tosoh G7 method in 2007-2008, Tosoh Corp).

For hormone analyses, the blood samples were processed in a centrifuge. Progesterone was measured by the immunofluorometric assay (Wallac, Finland) using Auto DELFIA kits; androstenedione, PRL, LH, and FSH, by the immunofluorometric assay; dehydroepiandrosterone sulfate (DHEAS), by radioimmunoassay (Cisbio International, France and DSL, Texas, USA); and insulin and 17-OHP, by radioimmunoassay using DSL kits. The testosterone and SHBG levels were measured using the electrochemiluminescent immunoassay (Modular, Roche). The free testosterone index was calculated based on the followed formula: total testosterone/SHBG*100. Free testosterone was calculated by Vermeulen's formula. All analyses were performed twice and the intra-assay and interassay coefficients of variation did not exceed 10% and 15%, respectively.

Endometrial biopsies Endometrial samples will be obtained using the Pipelle de Cornier catheter (Laboratoire CCD, Paris, France). Part of the material was embedded in paraffin for histomorphometric and immunohistochemical analyses, and the remainder was preserved in RNA for later molecular analyses.

Histochemistry Endometrial samples will be fixed for 24 hrs. in 10% formaldehyde, dehydrated in increasing concentrations of ethyl alcohol, cleared in xylene, and then embedded in paraffin. The paraffin-embedded samples will be then cut into ten 3-μm sections per subject. Eight of these sections were stained for Vascular Endothelial Growth Factor C (VEGF-C) and for immunohistochemistry (see below), and the two remaining sections will be stained with hematoxylin and eosin (H&E) to confirm the menstrual cycle phase using the criteria suggested by Noyes et al. (1953) and morphometry (see below).

Sections willl be dewaxed conventionally; 0.3% H2O2 will be used to inactivate endogenous peroxidase at room temperature for 10 min, followed by washing with distilled water three times. The sections were immersed in 0.01 M citrate buffer (pH 6.0) and then placed in a microwave oven for heating up to the boiling point. After 10 min, this process will be repeated twice; then, the sections were cooled at room temperature and washed twice with phosphate-buffered saline (PBS) (pH 7.4). A 5% bovine serum albumin (BSA) blocking solution was added at room temperature for 20, min and the excess liquid was discarded. Rabbit anti-human VEGF-C polyclonal antibodies (Cell Signaling, Danvers, MA, USA) (VEGF-C: diluted at 1:100) were added to the incubation at 37°C for 24 h, and the sections were then washed for 5 min. thrice. A biotinylated goat anti-rabbit IgG (Cell Signaling, Danvers, MA, USA) working solution will be added at 1:1000 dilution for incubation at 37°C for 20 min. After washing, SABC will be added to the incubation at 37°C for 20 min, followed by washing and color development via diaminobenzidine (DAB) (DAB color development kit, Dako, Dinamarca) at room temperature for 5 to 30 min., followed by washing with distilled water, haematoxylin re-staining dehydration via graded ethanol, transparency via xylene, sealing via neutral gum, and inspection under light microscope. The primary antibody was replaced with PBS as a negative control. The positive sections that stained satisfactorily in the pre-experiment were used as positive controls.

Morphological and histomorphometric analyses To quantify the parameters of interest, images were captured using a high-resolution camera (AxioCam-MCR, Carl Zeiss) adapted to a light microscope (Axiolab, Carl Zeiss) and adjusted with 40× objective lenses. The images were transmitted to a computer with AxioVision Rel 4.2 software (Carl Zeiss). For assessment of glandular and surface epithelial thickness, cell count, and counting newly formed blood vessels, ten images of each endometrial sample were made for each patient. For VEGF-C determination, the numerical density of blood vessels per mm2 will be established.

Statistical analyses The minimum sample size needed for each group will be determined from a pilot study with 10 women per group after pilot study. Thus, in calculating the sample size, the correlation between the group measurements will be considered. For the results of the number of endometrial glands, a type I error of 5% and a type II error of 20% (sample with 0.8% power) were adopted for the detection of >20% difference between groups. Commensurate with homogeneity, the quantitative data will be expressed as mean ± standard deviation. In conformity with data distribution, the Student t test or the Mann-Whitney U test will be used. The significance level was set at 95% (α ≤ 5%). Moreover, ANOVA or the Kruskal-Wallis test will be used for histologic and immunohistochemical comparisons, when the additional group (PCOS during the proliferative phase) was included. Then, in line with data distribution, either the Tukey test or the Dunn test will be applied. When possible, the subjects of Study A and B were combined for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Polycystic ovarian syndrome (defined by the Rotterdam criteria, which includes two of the following three features: a) oligo-amenorrhea; b) clinical or biochemical signs of hyperandrogenism; and c) polycystic ovaries) ages 18 to 35 years; must be able to swallow tables
2. Controls - the family planning outpatient office and healthy women ages 18 to 35 years with regular menstrual cycles, no evidence of hirsutism; must be able to swallow tables

Exclusion Criteria:: a) use of any hormone treatment in the previous 3 months; b) other causes of anovulation as evidenced by abnormal levels of prolactin, cortisol, dehydroepiandrosterone sulphate (DHEAS), 17-hydroxyprogesterone (17-OHP), androstenedione, thyroid-stimulating hormone (TSH), and free T4, in blood samples obtained between days 2 and 5 of the cycle in cycling subjects or on any other day in amenorrheic subjects; c) gynecologic disorders or other associated diseases, such as endometriosis, hypertension, or diabetes mellitus; d) follicle-stimulating hormone (FSH) >15 UI/L (cycle days 2-5); or e) a positive β-subunit of human chorionic gonadotropin (β-HCG); Clinical diagnosis of Alzheimer´s disease; ; insulin dependent diabetes; thryoid diasease.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2014-09-10 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
Endometrial biopsy | 3 months
  Number of patients with adequate changes of endometrium similar to luteal phase.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Hum Reprod. 2018 Sep 1;33(9):1602-1618. doi: 10.1093/humrep/dey256. PMID 30052961
- [Background] Azziz R, Carmina E, Dewailly D, Diamanti-Kandarakis E, Escobar-Morreale HF, Futterweit W, Janssen OE, Legro RS, Norman RJ, Taylor AE, Witchel SF; Androgen Excess Society. Positions statement: criteria for defining polycystic ovary syndrome as a predominantly hyperandrogenic syndrome: an Androgen Excess Society guideline. J Clin Endocrinol Metab. 2006 Nov;91(11):4237-45. doi: 10.1210/jc.2006-0178. Epub 2006 Aug 29. PMID 16940456
- [Background] Azziz R, Carmina E, Dewailly D, Diamanti-Kandarakis E, Escobar-Morreale HF, Futterweit W, Janssen OE, Legro RS, Norman RJ, Taylor AE, Witchel SF; Task Force on the Phenotype of the Polycystic Ovary Syndrome of The Androgen Excess and PCOS Society. The Androgen Excess and PCOS Society criteria for the polycystic ovary syndrome: the complete task force report. Fertil Steril. 2009 Feb;91(2):456-88. doi: 10.1016/j.fertnstert.2008.06.035. Epub 2008 Oct 23. PMID 18950759
- [Background] Trivax B, Azziz R. Diagnosis of polycystic ovary syndrome. Clin Obstet Gynecol. 2007 Mar;50(1):168-77. doi: 10.1097/GRF.0b013e31802f351b. PMID 17304034
- [Background] Giudice LC. Endometrium in PCOS: Implantation and predisposition to endocrine CA. Best Pract Res Clin Endocrinol Metab. 2006 Jun;20(2):235-44. doi: 10.1016/j.beem.2006.03.005. PMID 16772154
- [Background] Slayden OD, Nayak NR, Burton KA, Chwalisz K, Cameron ST, Critchley HO, Baird DT, Brenner RM. Progesterone antagonists increase androgen receptor expression in the rhesus macaque and human endometrium. J Clin Endocrinol Metab. 2001 Jun;86(6):2668-79. doi: 10.1210/jcem.86.6.7606. PMID 11397870
- [Background] Ochoa-Bernal MA, Fazleabas AT. Physiologic Events of Embryo Implantation and Decidualization in Human and Non-Human Primates. Int J Mol Sci. 2020 Mar 13;21(6):1973. doi: 10.3390/ijms21061973. PMID 32183093
- [Background] Sharpe A, Morley LC, Tang T, Norman RJ, Balen AH. Metformin for ovulation induction (excluding gonadotrophins) in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2019 Dec 17;12(12):CD013505. doi: 10.1002/14651858.CD013505. PMID 31845767
- [Background] Walls ML, Hunter T, Ryan JP, Keelan JA, Nathan E, Hart RJ. In vitro maturation as an alternative to standard in vitro fertilization for patients diagnosed with polycystic ovaries: a comparative analysis of fresh, frozen and cumulative cycle outcomes. Hum Reprod. 2015 Jan;30(1):88-96. doi: 10.1093/humrep/deu248. Epub 2014 Oct 29. PMID 25355587
- [Background] Simoes RS, Soares JM Jr, Simoes MJ, Nader HB, Baracat MCP, Maciel GAR, Serafini PC, Azziz R, Baracat EC. Small leucine-rich proteoglycans (SLRPs) in the endometrium of polycystic ovary syndrome women: a pilot study. J Ovarian Res. 2017 Aug 8;10(1):54. doi: 10.1186/s13048-017-0349-9. PMID 28789706
- [Background] Munro MG, Critchley HOD, Fraser IS; FIGO Menstrual Disorders Committee. The two FIGO systems for normal and abnormal uterine bleeding symptoms and classification of causes of abnormal uterine bleeding in the reproductive years: 2018 revisions. Int J Gynaecol Obstet. 2018 Dec;143(3):393-408. doi: 10.1002/ijgo.12666. Epub 2018 Oct 10. PMID 30198563
- [Background] Lai TH, Zhao Y, Shih IeM, Ho CL, Bankowski B, Vlahos N. Expression of L-selectin ligands in human endometrium during the implantation window after controlled ovarian stimulation for oocyte donation. Fertil Steril. 2006 Mar;85(3):761-3. doi: 10.1016/j.fertnstert.2005.08.023. PMID 16500358
- [Background] Quezada S, Avellaira C, Johnson MC, Gabler F, Fuentes A, Vega M. Evaluation of steroid receptors, coregulators, and molecules associated with uterine receptivity in secretory endometria from untreated women with polycystic ovary syndrome. Fertil Steril. 2006 Apr;85(4):1017-26. doi: 10.1016/j.fertnstert.2005.09.053. Epub 2006 Mar 9. PMID 16580389
- [Background] Qiao J, Wang L, Li R, Zhang X. Microarray evaluation of endometrial receptivity in Chinese women with polycystic ovary syndrome. Reprod Biomed Online. 2008 Sep;17(3):425-35. doi: 10.1016/s1472-6483(10)60228-3. PMID 18765015
- [Background] Amsterdam ESHRE/ASRM-Sponsored 3rd PCOS Consensus Workshop Group. Consensus on women's health aspects of polycystic ovary syndrome (PCOS). Hum Reprod. 2012 Jan;27(1):14-24. doi: 10.1093/humrep/der396. Epub 2011 Dec 5. PMID 22147920
- [Background] Griukova A, Deryabin P, Shatrova A, Burova E, Severino V, Farina A, Nikolsky N, Borodkina A. Molecular basis of senescence transmitting in the population of human endometrial stromal cells. Aging (Albany NY). 2019 Nov 5;11(21):9912-9931. doi: 10.18632/aging.102441. Epub 2019 Nov 5. PMID 31689238
- [Background] Apparao KB, Lovely LP, Gui Y, Lininger RA, Lessey BA. Elevated endometrial androgen receptor expression in women with polycystic ovarian syndrome. Biol Reprod. 2002 Feb;66(2):297-304. doi: 10.1095/biolreprod66.2.297. PMID 11804942
- [Background] Cheung AP. Ultrasound and menstrual history in predicting endometrial hyperplasia in polycystic ovary syndrome. Obstet Gynecol. 2001 Aug;98(2):325-31. doi: 10.1016/s0029-7844(01)01432-6. PMID 11506853
- [Background] Maliqueo M, Clementi M, Gabler F, Johnson MC, Palomino A, Sir-Petermann T, Vega M. Expression of steroid receptors and proteins related to apoptosis in endometria of women with polycystic ovary syndrome. Fertil Steril. 2003 Sep;80 Suppl 2:812-9. doi: 10.1016/s0015-0282(03)00987-7. PMID 14505758
- [Background] Heijnen EM, Eijkemans MJ, Hughes EG, Laven JS, Macklon NS, Fauser BC. A meta-analysis of outcomes of conventional IVF in women with polycystic ovary syndrome. Hum Reprod Update. 2006 Jan-Feb;12(1):13-21. doi: 10.1093/humupd/dmi036. Epub 2005 Aug 25. PMID 16123051
- [Result] Lopes IM, Baracat MC, Simoes Mde J, Simoes RS, Baracat EC, Soares JM Jr. Endometrium in women with polycystic ovary syndrome during the window of implantation. Rev Assoc Med Bras (1992). 2011 Nov-Dec;57(6):702-9. doi: 10.1590/s0104-42302011000600020. English, Portuguese. PMID 22249553
- [Result] de Medeiros SF, Yamamoto MMW, Souto de Medeiros MA, Barbosa BB, Soares JM, Baracat EC. Changes in clinical and biochemical characteristics of polycystic ovary syndrome with advancing age. Endocr Connect. 2020 Feb;9(2):74-89. doi: 10.1530/EC-19-0496. PMID 31905164
- [Result] Baracat MC, Serafini PC, Simoes Rdos S, Maciel GA, Soares JM Jr, Baracat EC. Systematic review of cell adhesion molecules and estrogen receptor expression in the endometrium of patients with polycystic ovary syndrome. Int J Gynaecol Obstet. 2015 Apr;129(1):1-4. doi: 10.1016/j.ijgo.2014.10.022. Epub 2014 Dec 18. PMID 25554522
- [Result] Lopes IM, Maganhin CC, Oliveira-Filho RM, Simoes RS, Simoes MJ, Iwata MC, Baracat EC, Soares JM Jr. Histomorphometric Analysis and Markers of Endometrial Receptivity Embryonic Implantation in Women With Polycystic Ovary Syndrome During the Treatment With Progesterone. Reprod Sci. 2014 Jul;21(7):930-938. doi: 10.1177/1933719113519169. Epub 2014 Jan 23. PMID 24458485
- [Result] Ejzenberg D, Simoes Mde J, Pinheiro W, Soares JM Junior, Serafini PC, Baracat EC. Blind aspiration biopsy versus a guided hysteroscopic technique for investigation of the endometrium in infertile women. Histol Histopathol. 2016 Sep;31(9):981-6. doi: 10.14670/HH-11-725. Epub 2016 Jan 25. PMID 26806353
- [Result] Ejzenberg D, Gomes TJO, Monteleone PAA, Serafini PC, Soares-Jr JM, Baracat EC. Prognostic factors for pregnancy after intrauterine insemination. Int J Gynaecol Obstet. 2019 Oct;147(1):65-72. doi: 10.1002/ijgo.12898. Epub 2019 Jul 23. PMID 31242330
- [Result] Savaris RF, Groll JM, Young SL, DeMayo FJ, Jeong JW, Hamilton AE, Giudice LC, Lessey BA. Progesterone resistance in PCOS endometrium: a microarray analysis in clomiphene citrate-treated and artificial menstrual cycles. J Clin Endocrinol Metab. 2011 Jun;96(6):1737-46. doi: 10.1210/jc.2010-2600. Epub 2011 Mar 16. PMID 21411543
- [Result] Giordano MV, Giordano LA, Gomes RC, Simoes RS, Nader HB, Giordano MG, Baracat EC, Soares Junior JM. The evaluation of endometrial sulfate glycosaminoglycans in women with polycystic ovary syndrome. Gynecol Endocrinol. 2015 Apr;31(4):278-81. doi: 10.3109/09513590.2014.989980. Epub 2014 Dec 1. PMID 25434369